CLINICAL TRIAL: NCT06803940
Title: Evaluation of Root Parallelism in Cases of Anterior Teeth Spacing Treated With Clear Aligner Versus Fixed Appliances
Brief Title: Evaluation of Root Parallelism in Cases of Anterior Teeth Spacing Clear Aligner Versus Fixed Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Amira Osama Elshall, Master's student, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-OR-23-09
Record Dates: First submitted 2025-01-05; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: The Present Study Aimed to Evaluate Root Parallelism in Cases of Anterior Teeth Spacing Treated With Clear Aligner Versus Fixed Orthodontic Appliances; Spacing Between Anterior Teeth
Keywords: Clear aligner, anterior spacing, root parallelism
MeSH Terms: interventions — Orthodontic Appliances, Removable; Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aligner (Experimental): intervention patient treated with clear aligner therapy
  Interventions: Procedure: clear aligner
- fixed appliance (Active Comparator): patient treated with conventional appliance
  Interventions: Procedure: orthodontic treatment

INTERVENTIONS:
Procedure: clear aligner — closing of spacing in anterior teeth with clear aligner therapy
  Arms: aligner
Procedure: orthodontic treatment — conventional fixed orthodontic appliance
  Arms: fixed appliance

SUMMARY:
evaluate root parallelism in cases of anterior teeth spacing treated with clear aligner versus fixed orthodontic appliances

ELIGIBILITY:
Inclusion Criteria: 1. Patients with anterior spacing as less than 2mm for anterior 2. Age range from 14 to 22 years old with no sex discrimination. 3. Good oral hygiene. 4. Presence of all permanent teeth not including third molars. 5. Provide informed consent and willingness to cooperate with study protocol.

Exclusion Criteria:

1. Medical problems or craniofacial disorders known to affect bone remodeling.
2. Congenital defect or deformed anterior teeth.
3. Presence of chronic or acute periodontal disease.
4. Radiographic evidence of bone loss.
5. History of systemic disease.
6. Previous orthodontic treatment.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
root parallelism | 6 months
  root angulation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: Undecided